CLINICAL TRIAL: NCT00158470
Title: Feasibility Study of a Once Daily Antiretroviral Regimen for HIV-Infected Patients With CD4 Below 200/mm3, in Hô Chi Minh City, Vietnam
Brief Title: Feasibility Study of a Once Daily Antiretroviral Regimen in Vietnam (ANRS 1210 VIETAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 1210 VIETAR; VIETAR
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infection
Keywords: HIV infection; injecting drug users; HAART; once daily regimen; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Didanosine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: efavirenz
Drug: didanosine
Drug: lamivudine

SUMMARY:
Access to care and treatment using antiretroviral drugs will be expanded in Vietnam in the next few years. The ANRS 1210 study is a pilot program to evaluate the feasibility of a simplified antiretroviral treatment using three antiretroviral drugs once a day. The objectives will be to assess the efficacy and the tolerance of this treatment and to better understand the difficulties linked to social and behavioural conditions of patients at different stages during the treatment.

DETAILED DESCRIPTION:
Despite a high number of infected subjects (estimated of 250,000 at the end of 2004) and a rapid spread of HIV infection in Vietnam, the use of anti-retroviral therapy remains limited. However, access to care and treatment will be expanded in Vietnam in the next few years with the support of national and international organisations. ANRS 1210 study is the first pilot program using highly active antiretroviral therapy (HAART) to evaluate the efficacy and the tolerance of an antiretroviral therapy delivered to adults in an external system of medical care, in Ho Chi Minh City. This feasibility study has also the objective to evaluate the cause of treatment failures and to assess social and behavioural conditions of patients at different stages during the treatment.

The present study is an open trial with direct individual benefit. The chosen treatment is a once-daily administration of 3TC, ddI and Efavirenz delivered to HIV infected adults with a CD4 count below 200/mm3. The duration of the study is eighteen months with a main evaluation at six months. One hundred patients will be selected in outpatient consultation of Binh Trieu hospital and Tropical Diseases Hospital of Ho Chi Minh City. The main criteria of evaluation will be the immunological response at 6 months, opportunistic infection events and the proportion of patients undergoing a regular monitoring at 6 months. Viral response will be also appreciated but, for technical question, will not be a main criteria of the study.

Patients are also administered a questionnaire by a trained independent interviewer about adherence to treatment, mental well-being, housing and nutrition, drug and sexual behaviour, social support and disclosure in order to study the associations between sociobehavioural dimensions, adherence and viral load at two successive follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old
* HIV infected
* Written informed consent signed
* CD4 count lower than 200/mm3
* No previous antiretroviral treatment
* Weight over 45 kilos and/or body mass index over 16
* Karnofsky Index over or equal to 70 percent

Exclusion Criteria:

* Pregnant woman or woman without effective contraception
* Opportunistic infection compromising the realisation of the treatment
* Tumoral pathology
* Progressive psychiatric affection
* Previous history of peripheral neuropathy or pancreatitis
* Hemoglobin above 90 g/l
* PMN neutrophil above 1.0G/l
* Platelets above 50G/l
* Liver enzymes over 5 times the normal values
* Lipase and/or amylase over 2 times the normal values
* Prothrombin rate above 50 percent
* Plasmatic creatinine over 200 micromoles/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
CD4 lymphocyte count after HAART | 6 months

SECONDARY OUTCOMES:
Evaluation of treatment failures causes | 12 months
Assessment of patients social and behavioral conditions at different stages during the treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves Follezou, Pr, Study Chair — CHU Pitié-Salpêtrière, Paris, France; Huu Chi Nguyen, Dr, Principal Investigator — Tropical Diseases Hospital - Ho Chi Minh City - Vietnam
Locations (2):
- Vietnam (2):
  - Binh Trieu Hospital, Ho Chi Minh City
  - Tropical Diseases Hospital, Ho Chi Minh City